CLINICAL TRIAL: NCT02536963
Title: Amblyopia and Strabismus Testing in Pediatrics
Brief Title: Improving Quality Vision Outcomes in Managed Care Setting While Reducing Cost by Use of Accurate, Automated Screening
Status: Completed | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: Kaiser Foundation Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: R44EY025926 (NIH)
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PVS Screening and reference examination: All enrolled participants will be screened with the Pediatric Vision Scanner (PVS screening) during a well-child visit to compare whether the results of the PVS match the results of the regular eye examination performed during the well-visit. They will then receive a reference examination performed by a fellowship-trained pediatric ophthalmologist. Results will be compared with PVS screening results.
  Interventions: Device: Pediatric Vision Scanning device; Other: Reference examination

INTERVENTIONS:
Device: Pediatric Vision Scanning device — The Pediatric Vision Scanner (PVS) performs a 3-second, non-invasive scan of both eyes simultaneously while a child looks at a single target. The scan will measure the frequency of the light waves that reflect off of the participants' eyes to determine the fixation state of the eye.
Other: Reference examination — Reference examination of the eyes will be performed by a fellowship-trained pediatric ophthalmologist.
  Other Names: Gold-standard eye exam

SUMMARY:
Amblyopia ("lazy eye") and strabismus (misaligned eyes) are medical eye conditions that combine as the leading causes of preventable vision loss in children. They are irreversible if not detected and corrected by the age of seven, however half of all cases are missed because the conditions do not always manifest themselves and pediatricians are unable to reliably detect the conditions. The current health care system badly needs an accurate and effective approach toward detecting amblyopia and strabismus in preschool children.

The study will be conducted in busy, ethnically and racially diverse primary care sites operated by the Kaiser Permanente system and compare the outcomes of testing with a Pediatric Vision Scanner with outcomes the current standard of care.

DETAILED DESCRIPTION:
After demonstrating feasibility, we will recruit 300 clinical trial participants during previously scheduled visits at two Kaiser Permanente of Southern California (KPSC) pediatric clinics. We will also send letters and placed phone calls to parents of eligible children who lived in cities proximal to the two clinics. Children will be considered eligible if age is ≥ 2 years old, less than 6 years old; have never visited an ophthalmologist (as this could indicate a pre-existing eye condition and/or introduce biased eye exam results if the physician had seen the patient before), are an active Kaiser Permanente member, and do not have a cognitive and/or developmental disability (ICD-10 codes Z82.79 and F84.0).

Interested participants will either visit an on-site ophthalmology clinic immediately following their pediatric visit or make a future appointment at one of two KPSC ophthalmology clinics. All study activities will be completed during one appointment. Research staff describe the study to parents and obtain informed consent, collected parent-reported demographic data about each participant, screen each participant using the PVS, and documented PVS results, test acquisition time, and participant cooperation. Testing will be performed in a dimly lit room with the child seated on a chair or parents lap. Per manufacturer recommendations, a background calibration measurement is first obtained off of the face with closed eyes. Then the child is asked to open both eyes and fixate on the smiley face target within the device while the binocular retinal polarization scan is performed. PVS results will be interpreted as either "pass" or "refer" based on manufacturer recommendations. Acquisition time is defined as time from when the research staff picked up the PVS to when the result is generated, and cooperation is defined as "excellent" or "fair" based on staff discretion (e.g., a patient who listens to instructions and completes the exam on the first try would be "excellent," whereas a patient who moves his/her head around during testing would be "fair"). A pediatric ophthalmologist masked to the PVS result then performs a gold standard eye examination. Possible gold standard examination results were "normal", "normal with risk factors" (Table Amblyopia Risk Factors - see protocol), "suspected binocular vision deficit," "suspected amblyopia," "amblyopia, "strabismus" and "amblyopia and strabismus." (Diagnostic Categories Rubric - see protocol). Results were mutually exclusive. To compare the PVS results to the gold standard eye examination among the 300 children eligible for analysis, we will perform a validation characteristics analysis with a 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-10, presenting for a well-visit (for enrollment for first primary outcome)
* Between the ages of 2-5, presenting for a well-visit (for enrollment for second primary outcome)

Exclusion Criteria:

* No developmental delay or cognitive deficit
* No visually obvious ocular conditions that would warrant specialist referral

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-5 who present themselves to the pediatric clinic for well-visits.
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Mehta, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Southern California Permanente Group, La Palma, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; cumulative results from the study may be presented in research journals and/or society conferences.

RESULTS

PARTICIPANT FLOW:
Groups:
- PVS Screening: All enrolled participants will be screened with the Pediatric Vision Scanner (PVS screening) during a well-child visit to compare whether the results of the PVS match the results of the regular eye examination performed during the well-visit.
  Pediatric Vision Scanning device: The Pediatric Vision Scanner (PVS) performs a 3-second, non-invasive scan of both eyes simultaneously while a child looks at a single target. The scan will measure the frequency of the light waves that reflect off of the participants' eyes to determine the fixation state of the eye.
  All enrolled participants will receive a reference examination performed by a fellowship-trained pediatric ophthalmologist. Results will be compared with PVS screening results.
  Reference examination: Reference examination of the eyes will be performed by a fellowship-trained pediatric ophthalmologist.
Period: Overall Study
Arm/Group | PVS Screening
Started | 318
Completed | 300
Not Completed | 18
Not completed — Withdrawal by Subject | 18

BASELINE CHARACTERISTICS:
Population: The participants who received the screening are the same participants who received the examination.
Groups:
- PVS Screening and Reference Examination: All enrolled participants will be screened with the Pediatric Vision Scanner (PVS screening) during a well-child visit to compare whether the results of the PVS match the results of the regular eye examination performed during the well-visit.
  Pediatric Vision Scanning device: The Pediatric Vision Scanner (PVS) performs a 3-second, non-invasive scan of both eyes simultaneously while a child looks at a single target. The scan will measure the frequency of the light waves that reflect off of the participants' eyes to determine the fixation state of the eye.
  All enrolled participants will receive a reference examination performed by a fellowship-trained pediatric ophthalmologist. Results will be compared with PVS screening results.
  Reference examination: Reference examination of the eyes will be performed by a fellowship-trained pediatric ophthalmologist.
Arm/Group | PVS Screening and Reference Examination
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 300
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 113
  Not Hispanic or Latino | 185
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 63
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 131
  More than one race | 70
  Unknown or Not Reported | 26
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: Detection of Amblyopia and Strabismus in Children Ages 2-5 Using Automated Pediatric Vision Scanner Device
Description: Screening device will provide a binocularity score from 0-100. Scores ≥60 indicate "normal" exams, while scores <60 are "refers" for amblyopia and strabismus. Device results will be compared to the gold standard eye examination performed by a pediatric ophthalmologist.
Time Frame: Screenings will be performed during a normally scheduled well-child visit, which lasts on average 20 minutes. Eye examinations for "refer" screenings will occur immediately after well-child visit.
Measure: Count of Participants; unit: Participants
Groups:
- PVS Screening and Reference Examination: All enrolled participants were screened with the Pediatric Vision Scanner (PVS screening) during a well-child visit to compare whether the results of the PVS match the results of the regular eye examination performed during the well-visit.
  Pediatric Vision Scanning device: The Pediatric Vision Scanner (PVS) performs a 3-second, non-invasive scan of both eyes simultaneously while a child looks at a single target. The scan will measure the frequency of the light waves that reflect off of the participants' eyes to determine the fixation state of the eye.
  All enrolled participants received a reference examination performed by a fellowship-trained pediatric ophthalmologist. Results will be compared with PVS screening results.
  Reference examination: Reference examination of the eyes will be performed by a fellowship-trained pediatric ophthalmologist.
Arm/Group | PVS Screening and Reference Examination
Number analyzed (Participants) | 300
Participants
  True positive - amblyopia with REFER result | 6
  True negative - control with PASS result | 249
  False negative - amblyopia with PASS result | 0
  False positive - control with REFER result | 45

ADVERSE EVENTS:
Time Frame: 1 day (date of data collection only)
Arm/Group | PVS Screening and Reference Examination
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02536963/ICF_000.pdf
  • Statistical Analysis Plan (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02536963/SAP_001.pdf
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02536963/Prot_002.pdf